CLINICAL TRIAL: NCT00232141
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multi-Center Trial of Pregabalin Versus Placebo in the Treatment of Neuropathic Pain Associated With HIV Neuropathy.
Brief Title: Study of Pregabalin Versus Placebo in the Treatment of Nerve Pain Associated With HIV Neuropathy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A0081066
Record Dates: First submitted 2005-09-30; First posted 2005-10-04 (Estimated); Results first posted 2009-08-11 (Estimated); Last update posted 2021-02-09 (Actual); Status verified 2009-06

CONDITIONS: HIV Infections; Peripheral Neuropathy
MeSH Terms: conditions — HIV Infections; Peripheral Nervous System Diseases | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: pregabalin
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: pregabalin — 75mg BID (can be titrated up to 150mg BID on day 4 based on individual response and up to 300mg BID at the end of week 1, visit 3 and end of week 2, visit 4)
  Arms: 1
Drug: Placebo — Placebo
  Arms: 2

SUMMARY:
Study to determine if pregabalin is more effective than placebo in treating subjects with nerve pain associated with HIV neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with confirmed diagnosis of HIV infection
* HIV-associated neuropathic pain (nerve pain) for at least 3 months prior to study start
* subjects with moderate to severe pain
* subjects on stable HIV and pain medications (some medications are not allowed to be taken while participating in the study).

Exclusion Criteria:

* Pregnant or breast feeding females
* subjects using street drugs or alcohol abusers during the study
* subject's on anti-diabetic medications
* use of neuroregenerative agents or neurotoxic chemotherapeutic agents 3 months prior to study start and throughout the study
* use of neurotoxic drugs (other than D-drugs) within a month prior to study start and throughout the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2005-10; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (34):
- United States (32):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Little Rock, Arkansas
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Sacramento, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, San Francisco, California
  - Pfizer Investigational Site, Stanford, California
  - Pfizer Investigational Site, West Hollywood, California
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Pensacola, Florida
  - Pfizer Investigational Site, Safety Harbor, Florida
  - Pfizer Investigational Site, Vero Beach, Florida
  - Pfizer Investigational Site, West Palm Beach, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Honolulu, Hawaii
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Springfield, Massachusetts
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Austin, Texas
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Longview, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Seattle, Washington
  - Pfizer Investigational Site, Milwaukee, Wisconsin
- Puerto Rico (2):
  - Pfizer Investigational Site, Ponce
  - Pfizer Investigational Site, San Juan

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081066&StudyName=Study%20of%20Pregabalin%20versus%20placebo%20in%20the%20treatment%20of%20Nerve%20Pain%20associated%20with%20HIV%20Neuropathy%20

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 43 centers in the United States; Study Initiation and Completion Dates: 6 October 2005 to 27 November 2007
Pre-assignment Details: A total of 472 subjects were screened for the study, and 302 subjects were randomized to study treatment.
Groups:
- Pregabalin: Study included a Screening phase, a 2-week double-blind Dose Adjustment phase, a 12-week double-blind Maintenance phase, and ended with a 1-week Taper/Follow-up phase. Subjects were randomized in a 1:1 ratio and were allowed to achieve a maximum dose of 600 mg/day (300 mg BID) and a minimum dose of 150 mg/day (75 mg BID) during the Maintenance phase.
- Placebo: Study included a Screening phase, a 2-week double-blind Dose Adjustment phase, a 12-week double-blind Maintenance phase, and ended with a 1-week Taper/Follow-up Phase. Subjects were randomized in a 1:1 ratio.
Period: Overall Study
Arm/Group | Pregabalin | Placebo
Started | 151 | 151
Completed | 120 | 125
Not Completed | 31 | 26
Not completed — Adverse Event | 9 | 4
Not completed — Lack of Efficacy | 0 | 3
Not completed — Lost to Follow-up | 9 | 6
Not completed — Other | 8 | 10
Not completed — Withdrawal by Subject | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pregabalin | Placebo | Total
Number analyzed (Participants) | 151 | 151 | 302
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.2 (8.1) | 46.8 (7.5) | 47.5 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 31 | 57
  Male | 125 | 120 | 245

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline for Numerical Rating Scale (NRS) Pain Scores at Endpoint-LOCF (Last Observation Carried Forward) Relative to Baseline
Description: Change from baseline in mean NRS-Pain scores at endpoint-LOCF. Daily pain scores were assessed on an 11-point numerical rating scale <(NRS)-Pain> ranging from 0 (no pain) to 10 (worst possible pain).
Time Frame: Baseline, Week 14
Population: ITT population (ie, full analysis set)=all randomized participants who took at least 1 dose & had at least 1 post-randomization efficacy assessment. The endpoint-LOCF mean value was computed from last 7 diary entries (Day 2 up to and including the day after the last dose w/n Dose-Adjustment or Maintenance phase (up to Day 99).
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 141 | 140
score on scale | -2.88 (0.21) | -2.63 (0.21)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Primary hypotheses : null (H0): µA=µP vs alternative (HA): µA≠µP (µA and µP represent true means for primary endpoint in active treatment & placebo groups respectively). Assumptions in power calculation: 2-sided test with type I error at α =0.05, type II error at β =0.10, & a common s.d of 2.2 for primary endpoint (based on previous clinical trial data). With n=150 subjects/ group (300 subjects overall) at least 90% power to detect a treatment difference of at least 1.1 in primary endpoint; Test type: Superiority or Other; p = 0.3914, ANCOVA — The analysis procedures planned will control the Type I error for the primary analysis. No multiplicity adjustment is needed for this two-group study; Mean Difference (Final Values) = -0.25, 95% CI [-0.83 to 0.32], Standard Error of Mean 0.29

2. Other Pre Specified Outcome: Change in NRS-Pain Scores From Baseline to Endpoint-BOCF (Modified Baseline Observation Carried Forward)
Description: Change from baseline in mean NRS-Pain scores at endpoint-BOCF. Daily pain scores were assessed on an 11-point numerical rating scale <(NRS)-Pain> ranging from 0 (no pain) to 10 (worst possible pain). Change from baseline in mean weekly pain scores was analyzed using longitudinal models assuming data were missing at random (MAR)
Time Frame: Baseline, Weeks 1 - 14 and Endpoint-BOCF
Population: ITT population; n = number of participants with data for analysis reported per week per treatment group (n=pregabalin, placebo).
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 141 | 140
score on scale
  Week 1 (n=136,133) | -1.14 (0.13) | -0.69 (0.13)
  Week 2 (n=126,132) | -1.92 (0.17) | -1.43 (0.17)
  Week 3 (n=118,121) | -2.36 (0.20) | -1.83 (0.20)
  Week 4 (n=118,124) | -2.66 (0.21) | -2.24 (0.20)
  Week 5 (n=116,121) | -2.79 (0.22) | -2.50 (0.21)
  Week 6 (n=111,119) | -2.98 (0.23) | -2.45 (0.22)
  Week 7 (n=112,111) | -3.22 (0.23) | -2.53 (0.23)
  Week 8 (n=111,111) | -3.33 (0.22) | -2.58 (0.22)
  Week 9 (n=107,111) | -3.09 (0.23) | -2.56 (0.23)
  Week 10 (n=106,114) | -2.98 (0.23) | -2.66 (0.22)
  Week 11 (n=102,106) | -3.05 (0.24) | -2.61 (0.24)
  Week 12 (n=96,105) | -3.14 (0.25) | -2.59 (0.24)
  Week 13 (n=96, 105) | -3.21 (0.25) | -2.59 (0.24)
  Week 14 (n=92,94) | -3.19 (0.26) | -2.70 (0.27)
  Endpoint BOCF (n=142,140) | -2.72 (0.21) | -2.64 (0.21)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 1; Test type: Superiority or Other; p = 0.0131, ANCOVA — All statistical tests of hypotheses were two-sided and at the 5% level of significance. All p-values for secondary or supportive analyses will be considered descriptive. No multiplicity adjustment was made for this two-group study; Mean Difference (Final Values) = -0.45, 95% CI [-0.81 to -0.10], Standard Error of Mean 0.18
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 2; Test type: Superiority or Other; p = 0.0393, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.49, 95% CI [-0.96 to -0.02], Standard Error of Mean 0.24
Statistical Analysis 3: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 3; Test type: Superiority or Other; p = 0.0554, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.54, 95% CI [-1.08 to 0.01], Standard Error of Mean 0.28
Statistical Analysis 4: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 4; Test type: Superiority or Other; p = 0.1513, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.42, 95% CI [-0.99 to 0.15], Standard Error of Mean 0.29
Statistical Analysis 5: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 5; Test type: Superiority or Other; p = 0.3345, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.29, 95% CI [-0.89 to 0.30], Standard Error of Mean 0.30
Statistical Analysis 6: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 6; Test type: Superiority or Other; p = 0.0879, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.53, 95% CI [-1.13 to 0.08], Standard Error of Mean 0.31
Statistical Analysis 7: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 7; Test type: Superiority or Other; p = 0.0307, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.69, 95% CI [-1.32 to -0.07], Standard Error of Mean 0.32
Statistical Analysis 8: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 8; Test type: Superiority or Other; p = 0.0156, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.75, 95% CI [-1.36 to -0.14], Standard Error of Mean 0.31
Statistical Analysis 9: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 9; Test type: Superiority or Other; p = 0.0981, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.53, 95% CI [-1.15 to 0.10], Standard Error of Mean 0.32
Statistical Analysis 10: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 10; Test type: Superiority or Other; p = 0.3060, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.32, 95% CI [-0.93 to 0.29], Standard Error of Mean 0.31
Statistical Analysis 11: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 11; Test type: Superiority or Other; p = 0.1874, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.43, 95% CI [-1.08 to 0.21], Standard Error of Mean 0.33
Statistical Analysis 12: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 12; Test type: Superiority or Other; p = 0.1025, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.56, 95% CI [-1.22 to 0.11], Standard Error of Mean 0.34
Statistical Analysis 13: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 13; Test type: Superiority or Other; p = 0.0662, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.63, 95% CI [-1.30 to 0.04], Standard Error of Mean 0.34
Statistical Analysis 14: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 14; Test type: Superiority or Other; p = 0.1856, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.49, 95% CI [-1.21 to 0.24], Standard Error of Mean 0.37
Statistical Analysis 15: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Endpoint; Test type: Superiority or Other; p = 0.7925, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.08, 95% CI [-0.66 to 0.50], Standard Error of Mean 0.30

3. Other Pre Specified Outcome: Responders- Decreases of at Least 50% in Mean Weekly Pain Score
Description: Number of subjects that experienced at least a 50% decrease in mean weekly pain.
Time Frame: Weeks 1-14 Endpoint BOCF (modified baseline observation carried forward)
Population: ITT population; n = number of participants with data for analysis reported per week per treatment group (n=pregabalin, placebo), BOCF = modified baseline observation carried forward
Measure: Number; unit: participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 146 | 147
participants
  Week 1 (n=140,141) | 13 | 6
  Week 2 (n=136,139) | 28 | 23
  Week 3 (n=131,133) | 35 | 33
  Week 4 (n=126,132) | 45 | 41
  Week 5 (n=124,131) | 48 | 47
  Week 6 (n=124,130) | 49 | 47
  Week 7 (n=125,124) | 53 | 38
  Week 8 (n=120,119) | 54 | 43
  Week 9 (n=116,121) | 50 | 45
  Week 10 (n=116,121) | 45 | 49
  Week 11 (n=113,117) | 43 | 46
  Week 12 (n=107,115) | 45 | 46
  Week 13 (n=103,111) | 45 | 47
  Week 14 (n=101,108) | 42 | 44
  Endpoint-BOCF (n=146,147) | 54 | 62
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 1; Test type: Superiority or Other; p = 0.1191, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Odds Ratio (OR) = 2.18, 95% CI [0.802 to 5.935]
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 2; Test type: Superiority or Other; p = 0.5041, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Odds Ratio (OR) = 1.24, 95% CI [0.666 to 2.301]
Statistical Analysis 3: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 3; Test type: Superiority or Other; p = 0.6859, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Odds Ratio (OR) = 1.13, 95% CI [0.638 to 1.985]
Statistical Analysis 4: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 4; Test type: Superiority or Other; p = 0.4140, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Odds Ratio (OR) = 1.25, 95% CI [0.735 to 2.116]
Statistical Analysis 5: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 5; Test type: Superiority or Other; p = 0.7852, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Odds Ratio (OR) = 1.07, 95% CI [0.644 to 1.794]
Statistical Analysis 6: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 6; Test type: Superiority or Other; p = 0.7399, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Odds Ratio (OR) = 1.09, 95% CI [0.654 to 1.817]
Statistical Analysis 7: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 7; Test type: Superiority or Other; p = 0.1055, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Odds Ratio (OR) = 1.57, 95% CI [0.913 to 2.701]
Statistical Analysis 8: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 8; Test type: Superiority or Other; p = 0.2107, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Odds Ratio (OR) = 1.41, 95% CI [0.829 to 2.401]
Statistical Analysis 9: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 9; Test type: Superiority or Other; p = 0.5270, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Odds Ratio (OR) = 1.19, 95% CI [0.697 to 2.046]
Statistical Analysis 10: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 10; Test type: Superiority or Other; p = 0.6845, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Odds Ratio (OR) = 0.89, 95% CI [0.513 to 1.546]
Statistical Analysis 11: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 11; Test type: Superiority or Other; p = 0.7737, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Odds Ratio (OR) = 0.92, 95% CI [0.522 to 1.619]
Statistical Analysis 12: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 12; Test type: Superiority or Other; p = 0.8853, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Odds Ratio (OR) = 1.04, 95% CI [0.597 to 1.818]
Statistical Analysis 13: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 13; Test type: Superiority or Other; p = 0.7712, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Odds Ratio (OR) = 1.09, 95% CI [0.612 to 1.946]
Statistical Analysis 14: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 14; Test type: Superiority or Other; p = 0.9586, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Odds Ratio (OR) = 1.02, 95% CI [0.574 to 1.796]
Statistical Analysis 15: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Endpoint-BOCF; Test type: Superiority or Other; p = 0.3482, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Odds Ratio (OR) = 0.79, 95% CI [0.486 to 1.283]

4. Other Pre Specified Outcome: Responders - Decreases of at Least 30% in Mean Weekly Pain Score
Description: Number of subjects that experienced at least 30% decrease in mean weekly pain.
Time Frame: Weeks 1-14 endpoint BOCF
Population: ITT population; n = number of participants with data for analysis reported per week per treatment group (n=pregabalin, placebo); BOCF = modified baseline observation carried forward
Measure: Number; unit: participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 146 | 147
participants
  Week 1 (n=140,141) | 33 | 21
  Week 2 (n=136,139) | 51 | 46
  Week 3 (n=131,133) | 63 | 51
  Week 4 (n=126,132) | 64 | 60
  Week 5 (n=124,131) | 65 | 68
  Week 6 (n=124,130) | 63 | 70
  Week 7 (n=125,124) | 69 | 64
  Week 8 (n=120,119) | 75 | 62
  Week 9 (n=116,121) | 68 | 65
  Week 10 (n=116,121) | 64 | 69
  Week 11 (n=113,117) | 67 | 63
  Week 12 (n=107,115) | 65 | 57
  Week 13 (n=103,111) | 62 | 62
  Week 14 (n=101,108) | 58 | 54
  Endpoint-BOCF (n=146,147) | 77 | 81
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 1; Test type: Superiority or Other; p = 0.1132, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Odds Ratio (OR) = 1.62, 95% CI [0.882 to 2.969]
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 2; Test type: Superiority or Other; p = 0.4687, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Odds Ratio (OR) = 1.20, 95% CI [0.731 to 1.978]
Statistical Analysis 3: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 3; Test type: Superiority or Other; p = 0.1546, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Odds Ratio (OR) = 1.44, 95% CI [0.877 to 2.375]
Statistical Analysis 4: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 4; Test type: Superiority or Other; p = 0.4216, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Odds Ratio (OR) = 1.23, 95% CI [0.7444 to 2.025]
Statistical Analysis 5: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 5; Test type: Superiority or Other; p = 0.7479, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Odds Ratio (OR) = 0.92, 95% CI [0.556 to 1.527]
Statistical Analysis 6: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 6; Test type: Superiority or Other; p = 0.3842, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Odds Ratio (OR) = 0.80, 95% CI [0.481 to 1.330]
Statistical Analysis 7: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 7; Test type: Superiority or Other; p = 0.8450, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Odds Ratio (OR) = 1.05, 95% CI [0.627 to 1.769]
Statistical Analysis 8: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 8; Test type: Superiority or Other; p = 0.1602, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Odds Ratio (OR) = 1.48, 95% CI [0.864 to 2.527]
Statistical Analysis 9: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 9; Test type: Superiority or Other; p = 0.6815, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Odds Ratio (OR) = 1.12, 95% CI [0.660 to 1.890]
Statistical Analysis 10: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 10; Test type: Superiority or Other; p = 0.5635, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Odds Ratio (OR) = 0.85, 95% CI [0.486 to 1.482]
Statistical Analysis 11: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 11; Test type: Superiority or Other; p = 0.4900, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Odds Ratio (OR) = 1.21, 95% CI [0.699 to 2.104]
Statistical Analysis 12: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 12; Test type: Superiority or Other; p = 0.1602, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Odds Ratio (OR) = 1.48, 95% CI [0.856 to 2.575]
Statistical Analysis 13: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 13; Test type: Superiority or Other; p = 0.5819, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Odds Ratio (OR) = 1.17, 95% CI [0.663 to 2.079]
Statistical Analysis 14: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 14; Test type: Superiority or Other; p = 0.2796, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Odds Ratio (OR) = 1.37, 95% CI [0.768 to 2.432]
Statistical Analysis 15: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Endpoint-BOCF; Test type: Superiority or Other; p = 0.5437, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Odds Ratio (OR) = 0.86, 95% CI [0.534 to 1.390]

5. Secondary Outcome: Change From Baseline for MOS (Medical Outcomes Study)-Sleep Subscales and Sleep Problem Indices
Description: Change from baseline in MOS-Sleep subscales & Sleep Problem Indices. Twelve item subject-rated questionnaire assessing sleep constructs. Scores range from 0 - 100 and higher scores reflect more impairment. Subscales "sleep adequacy", "quantity of sleep" and "optimal sleep" low scores reflect impairment.
Time Frame: Baseline, Week 14
Population: ITT Population; n = number of participants with data for analysis (n=pregabalin, placebo).
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 127 | 128
score on scale
  Disturbances (n=127,125) | -13.17 (1.82) | -14.71 (1.83)
  Quantity (n=123,122) | 0.39 (0.18) | 0.65 (0.19)
  Adequacy (n=126,128) | 10.04 (2.12) | 10.09 (2.11)
  Awaken Short of Breath or w/Headache (n=125,128) | -6.52 (1.82) | -7.93 (1.80)
  Somnolence (n=125,128) | -5.61 (1.81) | -7.01 (1.79)
  Snoring (n=122,126) | 4.34 (2.34) | -5.00 (2.29)
  Sleep problems Index I (n=122,127) | -10.11 (1.44) | -11.18 (1.41)
  Sleep problems Index II (n=122,125) | -10.16 (1.37) | -11.59 (1.35)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Disturbance; Test type: Superiority or Other; p = 0.5425, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 1.54, 95% CI [-3.44 to 6.52], Standard Error of Mean 2.53
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Quantity; Test type: Superiority or Other; p = 0.3184, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.25, 95% CI [-0.75 to 0.25], Standard Error of Mean 0.25
Statistical Analysis 3: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Adequacy; Test type: Superiority or Other; p = 0.9886, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.04, 95% CI [-5.81 to 5.72], Standard Error of Mean 2.92
Statistical Analysis 4: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Awaken Short of Breath or with Headache; Test type: Superiority or Other; p = 0.5742, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 1.41, 95% CI [-3.53 to 6.35], Standard Error of Mean 2.51
Statistical Analysis 5: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Somnolence; Test type: Superiority or Other; p = 0.5775, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 1.40, 95% CI [-3.54 to 6.33], Standard Error of Mean 2.50
Statistical Analysis 6: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Snoring; Test type: Superiority or Other; p = 0.0040, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 9.34, 95% CI [3.02 to 15.66], Standard Error of Mean 3.21
Statistical Analysis 7: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Sleep Problems Index I; Test type: Superiority or Other; p = 0.5882, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 1.07, 95% CI [-2.83 to 4.97], Standard Error of Mean 1.98
Statistical Analysis 8: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Sleep Problems Index II; Test type: Superiority or Other; p = 0.4516, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 1.42, 95% CI [-2.30 to 5.14], Standard Error of Mean 1.89

6. Secondary Outcome: Change From Baseline for Hospital Anxiety and Depression Scale (HADS) Subscales
Description: Change from Baseline in scale at endpoint: normal (score 0) to severe (score 21).
Time Frame: Baseline, Week 14
Population: ITT population
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 128 | 128
score on scale
  Anxiety | -1.33 (0.28) | -1.59 (0.28)
  Depression | -1.10 (0.26) | -1.52 (0.26)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Anxiety; Test type: Superiority or Other; p = 0.5105, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.26, 95% CI [-0.51 to 1.03], Standard Error of Mean 0.39
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Depression; Test type: Superiority or Other; p = 0.2513, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.42, 95% CI [-0.30 to 1.14], Standard Error of Mean 0.37

7. Secondary Outcome: Change From Baseline for Modified Brief Pain Inventory-Short Form (mBPI-sf) Scores
Description: Change from baseline to endpoint in the mBPI-sf to assess pain severity and pain interference with functional activities: 11-point scale ranging from "no pain" (0) to "pain as bad as you can imagine" (10)
Time Frame: Baseline, Week 14
Population: ITT Population; n = number of participants with data for analysis reported (n=pregabalin, placebo).
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 148 | 147
score on scale
  Pain Severity Index (n=148,147) | -2.42 (0.19) | -2.56 (0.19)
  Pain Interference Index (n=146,146) | -2.32 (0.18) | -2.39 (0.18)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Pain Severity Index; Test type: Superiority or Other; p = 0.5834, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.15, 95% CI [-0.38 to 0.67], Standard Error of Mean 0.27
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Pain Interference Index; Test type: Superiority or Other; p = 0.7783, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.07, 95% CI [-0.43 to 0.57], Standard Error of Mean 0.25

8. Secondary Outcome: Change From Baseline for NRS-Sleep Interference Scores
Description: 11-point numerical rating scale ranging from 0 (did not interfere with sleep) to 10 (completely interfered [unable to sleep due to pain])
Time Frame: Baseline, Week 14
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 140 | 140
score on scale | -2.53 (0.20) | -2.34 (0.20)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.4776, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.19, 95% CI [-0.73 to 0.34], Standard Error of Mean 0.27

9. Secondary Outcome: Categorized Patient Global Impression of Change (PGIC)
Description: The PGIC is a participant-rated instrument that measures change in the participants overall status on a 7-point scale. Scores range from 1 (very much improved) to 7 (very much worse). PGIC was evaluated using 3 categories of Improvement (Scores 1-3), No Change (Score 4), and Worsening (Scores 5-7).
Time Frame: Baseline, Week 14
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 149 | 150
participants
  Improved (scores 1-3) | 106 | 84
  No Change (score 4) | 17 | 32
  Worsened (scores 5-7) | 5 | 10
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.0077, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]

10. Secondary Outcome: Patient Global Impression of Change (PGIC) Rating
Description: PGIC is a participant-rated instrument that measures change in the participants overall status on a 7-point scale. Scores range from 1 (very much improved) to 7 (very much worse).
Time Frame: Baseline, Week 14, Endpoint-LOCF
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 149 | 150
participants
  Very much improved (score 1) | 27 | 27
  Much improved (score 2) | 41 | 38
  Minimally improved (score 3) | 38 | 19
  No change (score 4) | 17 | 32
  Minimally worse (score 5) | 2 | 5
  Much worse (score 6) | 3 | 5
  Very much worse (score 7) | 0 | 0
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.3852, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]

11. Secondary Outcome: Change in Neuropathic Pain Symptom Inventory (NPSI) Subscores and Total Intensity Scores
Description: Change in mean score NPSI, questionnaire evaluates symptoms of neuropathic pain. 10 pain descriptors questions answered on an 11-point scale 0 (no pain)-10 (most intense pain imaginable). 2 items related to temporal pain assessed on 5-point scales. The NPSI derives 5 pain subscores & a total intensity score calculated from the 5 pain subscores
Time Frame: Baseline, Week 14
Population: ITT Population; n = number of participants with data for analysis (n=pregabalin, placebo).
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 127 | 128
score on scale
  Burning (n=127,126) | -0.19 (0.02) | -0.22 (0.02)
  Pressing (n=125,126) | -0.17 (0.02) | -0.15 (0.02)
  Paroxysmal (n=127,127) | -0.16 (0.02) | -0.17 (0.02)
  Evoked (n=126,128) | -0.16 (0.02) | -0.15 (0.02)
  Paresthesia/dysesthesia (n=126,128) | -0.19 (0.02) | -0.23 (0.02)
  Total score (n=124,126) | -0.01 (0) | -0.01 (0)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Burning; Test type: Superiority or Other; p = 0.3097, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.03, 95% CI [-0.03 to 0.10], Standard Error of Mean 0.03
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Pressing; Test type: Superiority or Other; p = 0.6147, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.02, 95% CI [-0.07 to 0.04], Standard Error of Mean 0.03
Statistical Analysis 3: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Paroxysmal; Test type: Superiority or Other; p = 0.6838, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.01, 95% CI [-0.05 to 0.07], Standard Error of Mean 0.03
Statistical Analysis 4: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Evoked; Test type: Superiority or Other; p = 0.6479, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.01, 95% CI [-0.07 to 0.04], Standard Error of Mean 0.03
Statistical Analysis 5: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Paresthesia/dysesthesia; Test type: Superiority or Other; p = 0.1849, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.04, 95% CI [-0.02 to 0.11], Standard Error of Mean 0.03
Statistical Analysis 6: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Total Score; Test type: Superiority or Other; p = 0.5898, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0, 95% CI [0 to 0], Standard Error of Mean 0

12. Secondary Outcome: Change in Quantitative Assessment of Neuropathic Pain (QANeP)
Description: Change in a quantitative assessment of the participants' neuropathic pain were on an 11-point scale ranging from 0 (no pain) to 10 (most intense pain imaginable).
Time Frame: Baseline, Week 14
Population: ITT Population; n = number of participants with data for analysis (n=pregabalin, placebo).
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 120 | 119
score on scale
  Static mechanical allodynia (n=120,119) | -1.11 (0.21) | -1.22 (0.21)
  Dynamic mechanical allodynia (n=120,119) | -0.99 (0.18) | -0.77 (0.18)
  Punctate hyperalgesia testing area (n=118,119) | -0.78 (0.25) | -0.68 (0.26)
  Temporal summation to tactile stimuli (n=120,118) | -1.21 (0.24) | -1.04 (0.24)
  Cold allodynia testing area (n=120,117) | -1.19 (0.23) | -0.90 (0.24)
  Cold hyperalgesia testing area (n=117,112) | -0.82 (0.27) | -0.93 (0.28)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Static mechanical allodynia; Test type: Superiority or Other; p = 0.6865, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.12, 95% CI [-0.45 to 0.68], Standard Error of Mean 0.29
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Dynamic mechanical allodynia; Test type: Superiority or Other; p = 0.3787, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.22, 95% CI [-0.71 to 0.27], Standard Error of Mean 0.25
Statistical Analysis 3: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Punctate hyperalgesia testing area; Test type: Superiority or Other; p = 0.7704, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.10, 95% CI [-0.79 to 0.59], Standard Error of Mean 0.35
Statistical Analysis 4: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Temporal summation to tactile stimuli; Test type: Superiority or Other; p = 0.6088, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.17, 95% CI [-0.82 to 0.48], Standard Error of Mean 0.33
Statistical Analysis 5: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Cold allodynia testing area; Test type: Superiority or Other; p = 0.3767, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.29, 95% CI [-0.93 to 0.35], Standard Error of Mean 0.33
Statistical Analysis 6: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Cold hyperalgesia testing area; Test type: Superiority or Other; p = 0.7689, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.11, 95% CI [-0.64 to 0.86], Standard Error of Mean 0.38

13. Other Pre Specified Outcome: Duration Adjusted Average Change From Baseline in NRS Pain Scores
Description: Duration Adjusted Average Change(DAAC) in NRS-Pain score = (mean at observation - mean at baseline)x(proportion of planned study duration that the subject completed).
Time Frame: Weekly: Week 1 - Week 14
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 141 | 140
score on scale | -2.45 (0.18) | -2.07 (0.18)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.1277, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.38, 95% CI [-0.86 to 0.11], Standard Error of Mean 0.25

14. Secondary Outcome: Change in NRS-Sleep Interference Scores
Description: Change in mean Pain-related sleep interference was assessed on an 11-point scale from 0 (did not interfere with sleep) to 10 (completely interfered [unable to sleep due to pain]). Weekly mean score was the sum of the daily diary scores divided by the number of diary entries during that week.
Time Frame: Baseline, Weeks 1-14
Population: ITT Population; n = number of participants with data for analysis (n=pregabalin, placebo).
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 135 | 133
score on scale
  Week 1 (n=135, 133) | -1.04 (0.13) | -0.68 (0.13)
  Week 2 (n=123,132) | -1.99 (0.17) | -1.36 (0.16)
  Week 3 (n=117,121) | -2.26 (0.19) | -1.68 (0.19)
  Week 4 (n=117,124) | -2.34 (0.20) | -2.01 (0.19)
  Week 5 (n=115,121) | -2.57 (0.20) | -2.22 (0.19)
  Week 6 (n=110,119) | -2.73 (0.20) | -2.18 (0.19)
  Week 7 (n=110,111) | -2.89 (0.21) | -2.28 (0.21)
  Week 8 (n=109,111) | -2.98 (0.21) | -2.29 (0.21)
  Week 9 (n=105,111) | -2.73 (0.22) | -2.25 (0.21)
  Week 10 (n=104,114) | -2.79 (0.22) | -2.32 (0.20)
  Week 11 (n=100,106) | -2.76 (0.22) | -2.32 (0.21)
  Week 12 (n=94,105) | -2.83 (0.24) | -2.29 (0.22)
  Week 13 (n=94,105) | -2.95 (0.24) | -2.28 (0.22)
  Week 14 (n=90,94) | -2.93 (0.25) | -2.30 (0.25)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 1; Test type: Superiority or Other; p = 0.0469, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.36, 95% CI [-0.71 to -0.00], Standard Error of Mean 0.18
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 2; Test type: Superiority or Other; p = 0.0067, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.63, 95% CI [-1.08 to -0.18], Standard Error of Mean 0.23
Statistical Analysis 3: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 3; Test type: Superiority or Other; p = 0.0310, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.58, 95% CI [-1.10 to -0.05], Standard Error of Mean 0.27
Statistical Analysis 4: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 4; Test type: Superiority or Other; p = 0.2088, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.34, 95% CI [-0.86 to 0.19], Standard Error of Mean 0.27
Statistical Analysis 5: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 5; Test type: Superiority or Other; p = 0.1849, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.35, 95% CI [-0.87 to 0.17], Standard Error of Mean 0.26
Statistical Analysis 6: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 6; Test type: Superiority or Other; p = 0.0452, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.55, 95% CI [-1.09 to -0.01], Standard Error of Mean 0.27
Statistical Analysis 7: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 7; Test type: Superiority or Other; p = 0.0359, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.61, 95% CI [-1.18 to -0.04], Standard Error of Mean 0.29
Statistical Analysis 8: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 8; Test type: Superiority or Other; p = 0.0184, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.69, 95% CI [-1.26 to -0.12], Standard Error of Mean 0.29
Statistical Analysis 9: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 9; Test type: Superiority or Other; p = 0.1043, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.48, 95% CI [-1.06 to 0.10], Standard Error of Mean 0.29
Statistical Analysis 10: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 10; Test type: Superiority or Other; p = 0.1053, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.47, 95% CI [-1.04 to 0.10], Standard Error of Mean 0.29
Statistical Analysis 11: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 11; Test type: Superiority or Other; p = 0.1440, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.44, 95% CI [-1.03 to 0.15], Standard Error of Mean 0.30
Statistical Analysis 12: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 12; Test type: Superiority or Other; p = 0.0866, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.55, 95% CI [-1.17 to 0.08], Standard Error of Mean 0.32
Statistical Analysis 13: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 13; Test type: Superiority or Other; p = 0.0359, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.67, 95% CI [-1.30 to -0.04], Standard Error of Mean 0.32
Statistical Analysis 14: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 14; Test type: Superiority or Other; p = 0.0711, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.62, 95% CI [-1.30 to 0.05], Standard Error of Mean 0.34

15. Secondary Outcome: Shift in Hospital Anxiety and Depression (HADS) Subscales
Description: Anxiety subscale analyzes generalized anxiety (anxious mood,restlessness, anxious thoughts, panic attacks). The depression subscale focuses on the state of lost interest and diminished pleasure response. A score of Normal = 0-7, Mild = 8-10, Moderate = 11-14, Severe = 15-21.
Time Frame: Baseline, Week 14
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 128 | 128
participants
  Anxiety-normal (baseline&endpoint) | 47 | 55
  Anxiety-normal (baseline)& mild (endpoint) | 7 | 6
  Anxiety-normal (baseline)& moderate(endpoint) | 2 | 2
  Anxiety-normal(baseline)&severe(endpoint) | 0 | 0
  Anxiety-mild(baseline)& normal(endpoint) | 23 | 19
  Anxiety-mild(baseline)& mild(endpoint) | 7 | 6
  Anxiety-mild(baseline)& moderate(endpoint) | 2 | 6
  Anxiety-mild(baseline)& severe(endpoint) | 2 | 0
  Anxiety-moderate(baseline)& normal(endpoint) | 11 | 8
  Anxiety-moderate(baseline)& mild(endpoint) | 6 | 9
  Anxiety-moderate(baseline)& moderate(endpoint) | 8 | 5
  Anxiety-moderate(baseline)& severe(endpoint) | 3 | 1
  Anxiety-severe(baseline)& normal(endpoint) | 0 | 1
  Anxiety-severe(baseline)& mild(endpoint) | 1 | 2
  Anxiety-severe(baseline)& moderate(endpoint) | 7 | 6
  Anxiety-severe(baseline)&severe(endpoint) | 2 | 2
  Depression-normal (baseline&endpoint) | 75 | 69
  Depression-normal (baseline)&mild (endpoint) | 8 | 7
  Depression-normal (baseline)&moderate (endpoint) | 2 | 2
  Depression-normal (baseline)&severe (endpoint) | 1 | 0
  Depression-mild (baseline)&normal(endpoint) | 19 | 21
  Depression-mild (baseline)&mild(endpoint) | 5 | 5
  Depression-mild (baseline)&moderate(endpoint) | 3 | 2
  Depression-mild (baseline)&severe(endpoint) | 0 | 0
  Depression-moderate (baseline)&normal(endpoint) | 5 | 11
  Depression-moderate (baseline)&mild(endpoint) | 6 | 7
  Depression-moderate (baseline)&moderate(endpoint) | 2 | 2
  Depression-moderate (baseline)&severe(endpoint) | 1 | 1
  Depression-severe (baseline)&normal(endpoint) | 0 | 0
  Depression-severe (baseline)&mild(endpoint) | 0 | 0
  Depression-severe (baseline)&moderate(endpoint) | 0 | 0
  Depression-severe (baseline)&severe(endpoint) | 1 | 1

16. Secondary Outcome: Change in Brief Pain Inventory-short Form (BPI-sf) Scores (The Worst Pain in the Past 24 Hours)
Description: Change in mean BPI-sf, is a self-administered questionnaire to assess pain severity 0 (no pain to 10 (pain as bad as you can imagine) and pain interference 0 (does not interfere) to 10 (completely interferes) during a 24 hour period. The BPI-sf was used to derive the change from baseline in 4 pain severity questions & 7 pain interference questions.
Time Frame: Baseline, Weeks 1,2,6,10,14, Endpoint - LOCF
Population: ITT population; n = number of participants with data for analysis (n=pregabalin, placebo).
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 148 | 147
score on scale
  Week 1 (n=145,147) | -1.52 (0.17) | -1.09 (0.17)
  Week 2 (n=139,143) | -2.18 (0.20) | -2.20 (0.20)
  Week 6 (n=132,134) | -3.08 (0.21) | -2.95 (0.21)
  Week 10 (n=126,128) | -3.02 (0.21) | -3.03 (0.21)
  Week 14 (n=116,120) | -2.97 (0.24) | -3.01 (0.24)
  Endpoint -LOCF (n=148,147) | -2.82 (0.22) | -2.88 (0.22)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 1; Test type: Superiority or Other; p = 0.0685, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.43, 95% CI [-0.89 to 0.03], Standard Error of Mean 0.23
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 2; Test type: Superiority or Other; p = 0.9280, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.03, 95% CI [-0.52 to 0.57], Standard Error of Mean 0.28
Statistical Analysis 3: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 6; Test type: Superiority or Other; p = 0.6672, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.13, 95% CI [-0.71 to 0.45], Standard Error of Mean 0.29
Statistical Analysis 4: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 10; Test type: Superiority or Other; p = 0.9731, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.01, 95% CI [-0.57 to 0.59], Standard Error of Mean 0.29
Statistical Analysis 5: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 14; Test type: Superiority or Other; p = 0.9045, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.04, 95% CI [-0.61 to 0.69], Standard Error of Mean 0.33
Statistical Analysis 6: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Endpoint; Test type: Superiority or Other; p = 0.8298, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.07, 95% CI [-0.53 to 0.66], Standard Error of Mean 0.30

17. Secondary Outcome: Change in Brief Pain Inventory-sf Scores (The Least Pain in the Past 24 Hours)
Description: as for outcome 16
Time Frame: Baseline, Weeks 1,2,6,10,14, Endpoint-LOCF
Population: ITT population; n = number of participants with data for analysis (n=pregabalin, placebo).
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 148 | 147
score on scale
  Week 1 (n=145,147) | -0.84 (0.18) | -0.80 (0.17)
  Week 2 (n=139,143) | -1.49 (0.19) | -1.44 (0.19)
  Week 6 (n=132,134) | -2.37 (0.19) | -2.05 (0.18)
  Week 10 (n=126,128) | -2.32 (0.20) | -2.13 (0.19)
  Week 14 (n=116,120) | -2.27 (0.20) | -2.41 (0.20)
  Endpoint (n=148,147) | -2.07 (0.19) | -2.20 (0.19)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 1; Test type: Superiority or Other; p = 0.8605, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.04, 95% CI [-0.52 to 0.44], Standard Error of Mean 0.24
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 2; Test type: Superiority or Other; p = 0.8348, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.06, 95% CI [-0.58 to 0.47], Standard Error of Mean 0.27
Statistical Analysis 3: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 6; Test type: Superiority or Other; p = 0.2227, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.32, 95% CI [-0.83 to 0.19], Standard Error of Mean 0.26
Statistical Analysis 4: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 10; Test type: Superiority or Other; p = 0.4753, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.19, 95% CI [-0.73 to 0.34], Standard Error of Mean 0.27
Statistical Analysis 5: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 14; Test type: Superiority or Other; p = 0.6017, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.14, 95% CI [-0.40 to 0.68], Standard Error of Mean 0.27
Statistical Analysis 6: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Endpoint; Test type: Superiority or Other; p = 0.6158, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.13, 95% CI [-0.38 to 0.64], Standard Error of Mean 0.26

18. Secondary Outcome: Change in Brief Pain Inventory-sf Scores (Average Level of Pain in the Past 24 Hours)
Description: as for outcome 16
Time Frame: Baseline, Weeks 1,2,6,10,14 and Endpoint
Population: ITT population; n = number of participants with data for analysis (n=pregabalin, placebo).
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 148 | 147
score on scale
  Week 1 (n=145,147) | -1.15 (0.16) | -0.90 (0.16)
  Week 2 (n=139,143) | -1.79 (0.17) | -1.77 (0.17)
  Week 6 (n=132,134) | -2.64 (0.20) | -2.55 (0.19)
  Week 10 (n=126,128) | -2.86 (0.20) | -2.61 (0.19)
  Week 14 (n=116,120) | -2.58 (0.22) | -2.71 (0.22)
  Endpoint (n=148,147) | -2.37 (0.20) | -2.60 (0.20)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 1; Test type: Superiority or Other; p = 0.2390, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.26, 95% CI [-0.69 to 0.17], Standard Error of Mean 0.22
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 2; Test type: Superiority or Other; p = 0.9444, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.02, 95% CI [-0.49 to 0.45], Standard Error of Mean 0.24
Statistical Analysis 3: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 6; Test type: Superiority or Other; p = 0.7386, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.09, 95% CI [-0.63 to 0.45], Standard Error of Mean 0.27
Statistical Analysis 4: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 10; Test type: Superiority or Other; p = 0.3493, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.25, 95% CI [-0.79 to 0.28], Standard Error of Mean 0.27
Statistical Analysis 5: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 14; Test type: Superiority or Other; p = 0.6596, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.13, 95% CI [-0.46 to 0.73], Standard Error of Mean 0.30
Statistical Analysis 6: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Endpoint; Test type: Superiority or Other; p = 0.4075, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.23, 95% CI [-0.31 to 0.77], Standard Error of Mean 0.27

19. Secondary Outcome: Change in Brief Pain Inventory-sf Scores (How Much Pain Are You Having Right Now)
Description: as for outcome 16
Time Frame: Baseline, Weeks 1,2,6,10,14 and Endpoint
Population: ITT population; n = number of participants with data for analysis (n=pregabalin, placebo).
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 148 | 147
score on scale
  Week 1 (n=144,147) | -1.56 (0.17) | -1.01 (0.17)
  Week 2 (n=139,143) | -2.02 (0.19) | -1.98 (0.19)
  Week 6 (n=132,134) | -2.66 (0.20) | -2.66 (0.20)
  Week 10 (n=126,128) | -2.72 (0.20) | -2.57 (0.20)
  Week 14 (n=116, 120) | -2.43 (0.23) | -2.72 (0.22)
  Endpoint (n=148,147) | -2.26 (0.21) | -2.57 (0.21)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 1; Test type: Superiority or Other; p = 0.0202, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.55, 95% CI [-1.01 to -0.09], Standard Error of Mean 0.23
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 2; Test type: Superiority or Other; p = 0.8865, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.04, 95% CI [-0.55 to 0.47], Standard Error of Mean 0.26
Statistical Analysis 3: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 6; Test type: Superiority or Other; p = 0.9964, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.00, 95% CI [-0.54 to 0.54], Standard Error of Mean 0.27
Statistical Analysis 4: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 10; Test type: Superiority or Other; p = 0.5993, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.15, 95% CI [-0.70 to 0.41], Standard Error of Mean 0.28
Statistical Analysis 5: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 14; Test type: Superiority or Other; p = 0.3553, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.29, 95% CI [-0.33 to 0.90], Standard Error of Mean 0.31
Statistical Analysis 6: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Endpoint; Test type: Superiority or Other; p = 0.2771, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.31, 95% CI [-0.25 to 0.88], Standard Error of Mean 0.29

20. Secondary Outcome: Change in Brief Pain Inventory-sf Scores (During the Past 24 Hours, How Pain Has Interfered With Your General Activity)
Description: as for outcome 16
Time Frame: Baseline, Weeks 1,2,6,10,14 and Endpoint
Population: ITT population; n = number of participants with data for analysis (n=pregabalin, placebo).
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 148 | 147
score on scale
  Week 1 (n=145,147) | -1.35 (0.19) | -1.04 (0.19)
  Week 2 (n=139,143) | -1.95 (0.19) | -1.87 (0.19)
  Week 6 (n=132,134) | -2.37 (0.19) | -2.25 (0.19)
  Week 10 (n=125,128) | -2.32 (0.19) | -2.26 (0.19)
  Week 14 (n=116,120) | -2.16 (0.22) | -2.46 (0.21)
  Endpoint (n=148,147) | -2.15 (0.20) | -2.23 (0.20)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 1; Test type: Superiority or Other; p = 0.2352, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.31, 95% CI [-0.82 to 0.20], Standard Error of Mean 0.26
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 2; Test type: Superiority or Other; p = 0.7607, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.08, 95% CI [-0.60 to 0.44], Standard Error of Mean 0.26
Statistical Analysis 3: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 6; Test type: Superiority or Other; p = 0.6563, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.12, 95% CI [-0.64 to 0.40], Standard Error of Mean 0.27
Statistical Analysis 4: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 10; Test type: Superiority or Other; p = 0.8319, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.06, 95% CI [-0.58 to 0.47], Standard Error of Mean 0.27
Statistical Analysis 5: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 14; Test type: Superiority or Other; p = 0.3086, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.30, 95% CI [-0.28 to 0.89], Standard Error of Mean 0.30
Statistical Analysis 6: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Endpoint; Test type: Superiority or Other; p = 0.7972, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.07, 95% CI [-0.48 to 0.62], Standard Error of Mean 0.28

21. Secondary Outcome: Change in Brief Pain Inventory-sf Scores (During the Past 24 Hours, How Pain Has Interfered With Your Mood)
Description: as for outcome 16
Time Frame: Baseline, Weeks 1,2,6,10,14 and Endpoint
Population: ITT population; n = number of participants with data for analysis (n=pregabalin, placebo).
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 147 | 147
score on scale
  Week 1 (n=144,147) | -1.58 (0.21) | -1.20 (0.20)
  Week 2 (n=138,143) | -2.23 (0.23) | -2.06 (0.22)
  Week 6 (n=131,134) | -2.60 (0.20) | -2.41 (0.20)
  Week 10 (n=125,128) | -2.52 (0.20) | -2.37 (0.20)
  Week 14 (n=115,120) | -2.53 (0.22) | -2.76 (0.21)
  Endpoint (n=147,147) | -2.31 (0.20) | -2.46 (0.20)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 1; Test type: Superiority or Other; p = 0.1863, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.38, 95% CI [-0.94 to 0.18], Standard Error of Mean 0.28
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 2; Test type: Superiority or Other; p = 0.5953, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.16, 95% CI [-0.77 to 0.44], Standard Error of Mean -0.31
Statistical Analysis 3: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 6; Test type: Superiority or Other; p = 0.5080, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.18, 95% CI [-0.73 to 0.36], Standard Error of Mean 0.28
Statistical Analysis 4: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 10; Test type: Superiority or Other; p = 0.5842, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.15, 95% CI [-0.70 to 0.39], Standard Error of Mean 0.28
Statistical Analysis 5: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 14; Test type: Superiority or Other; p = 0.4286, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.24, 95% CI [-0.35 to 0.83], Standard Error of Mean 0.30
Statistical Analysis 6: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Endpoint; Test type: Superiority or Other; p = 0.5766, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.16, 95% CI [-0.40 to 0.71], Standard Error of Mean 0.28

22. Secondary Outcome: Change in Brief Pain Inventory-sf Scores (During the Past 24 Hours, How Pain Has Interfered With Your Walking Ability)
Description: as for outcome 16
Time Frame: Baseline, Weeks 1,2,6,10,14 and Endpoint
Population: ITT population; n = number of participants with data for analysis (n=pregabalin, placebo).
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 148 | 147
score on scale
  Week 1 (n=144,147) | -1.40 (0.21) | -1.23 (0.20)
  Week 2 (n=139,142) | -1.84 (0.22) | -1.84 (0.21)
  Week 6 (n=132,134) | -2.44 (0.21) | -2.33 (0.20)
  Week 10 (n=125,128) | -2.13 (0.20) | -2.33 (0.20)
  Week 14 (n=115,120) | -2.09 (0.22) | -2.54 (0.22)
  Endpoint (n=148,147) | -2.11 (0.21) | -2.42 (0.21)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 1; Test type: Superiority or Other; p = 0.5493, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.17, 95% CI [-0.73 to 0.39], Standard Error of Mean 0.28
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 2; Test type: Superiority or Other; p = 0.9875, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.00, 95% CI [-0.58 to 0.59], Standard Error of Mean 0.30
Statistical Analysis 3: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 6; Test type: Superiority or Other; p = 0.6931, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.11, 95% CI [-0.68 to 0.45], Standard Error of Mean 0.29
Statistical Analysis 4: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 10; Test type: Superiority or Other; p = 0.4614, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.20, 95% CI [-0.34 to 0.75], Standard Error of Mean 0.28
Statistical Analysis 5: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 14; Test type: Superiority or Other; p = 0.1467, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.45, 95% CI [-0.16 to 1.06], Standard Error of Mean 0.31
Statistical Analysis 6: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Endpoint; Test type: Superiority or Other; p = 0.2819, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.31, 95% CI [-0.25 to 0.87], Standard Error of Mean 0.29

23. Secondary Outcome: Change in Brief Pain Inventory-sf Scores (During the Past 24 Hours, How Pain Has Interfered With Your Normal Work Including Both Work Outside the Home and Housework)
Description: as for outcome 16
Time Frame: Baseline, Weeks 1,2,6,10,14 and Endpoint
Population: ITT population; n = number of participants with data for analysis (n=pregabalin, placebo).
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 147 | 147
score on scale
  Week 1 (n=144,147) | -1.47 (0.19) | -1.42 (0.18)
  Week 2 (n=138,143) | -2.10 (0.20) | -1.99 (0.20)
  Week 6 (n=130,134) | -2.54 (0.19) | -2.45 (0.19)
  Week 10 (n=125,128) | -2.49 (0.20) | -2.36 (0.20)
  Week 14 (n=114,120) | -2.21 (0.23) | -2.70 (0.22)
  Endpoint (n=147,147) | -2.30 (0.20) | -2.61 (0.20)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 1; Test type: Superiority or Other; p = 0.8727, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.04, 95% CI [-0.55 to 0.46], Standard Error of Mean 0.26
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 2; Test type: Superiority or Other; p = 0.6897, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.11, 95% CI [-0.65 to 0.43], Standard Error of Mean 0.28
Statistical Analysis 3: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 6; Test type: Superiority or Other; p = 0.7527, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.08, 95% CI [-0.60 to 0.44], Standard Error of Mean 0.26
Statistical Analysis 4: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 10; Test type: Superiority or Other; p = 0.6394, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.13, 95% CI [-0.67 to 0.41], Standard Error of Mean 0.28
Statistical Analysis 5: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 14; Test type: Superiority or Other; p = 0.1188, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.49, 95% CI [-0.13 to 1.11], Standard Error of Mean 0.31
Statistical Analysis 6: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Endpoint; Test type: Superiority or Other; p = 0.2685, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.31, 95% CI [-0.24 to 0.87], Standard Error of Mean 0.28

24. Secondary Outcome: Change in Brief Pain Inventory-sf Scores (During the Past 24 Hours, How Pain Has Interfered With Your Relations With Other People)
Description: as for outcome 16
Time Frame: Baseline, Weeks 1,2,6,10,14 and Endpoint
Population: ITT population; n = number of participants with data for analysis (n=pregabalin, placebo).
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 148 | 147
score on scale
  Week 1 (n=145,147) | -1.06 (0.21) | -0.87 (0.20)
  Week 2 (n=139,143) | -1.54 (0.22) | -1.39 (0.21)
  Week 6 (n=132,134) | -1.91 (0.19) | -1.67 (0.19)
  Week 10 (n=126,128) | -1.84 (0.19) | -1.91 (0.19)
  Week 14 (n=115,120) | -2.08 (0.20) | -2.10 (0.19)
  Endpoint (n=148,147) | -2.00 (0.19) | -1.99 (0.19)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 1; Test type: Superiority or Other; p = 0.4991, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.19, 95% CI [-0.74 to 0.36], Standard Error of Mean 0.28
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 2; Test type: Superiority or Other; p = 0.6094, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.15, 95% CI [-0.73 to 0.43], Standard Error of Mean 0.30
Statistical Analysis 3: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 6; Test type: Superiority or Other; p = 0.3669, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.24, 95% CI [-0.76 to 0.28], Standard Error of Mean 0.26
Statistical Analysis 4: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 10; Test type: Superiority or Other; p = 0.7641, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.08, 95% CI [-0.43 to 0.59], Standard Error of Mean 0.26
Statistical Analysis 5: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 14; Test type: Superiority or Other; p = 0.9428, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.02, 95% CI [-0.51 to 0.55], Standard Error of Mean 0.27
Statistical Analysis 6: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Endpoint; Test type: Superiority or Other; p = 0.9508, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.02, 95% CI [-0.52 to 0.49], Standard Error of Mean 0.26

25. Secondary Outcome: Change in Brief Pain Inventory-sf Scores (During the Past 24 Hours, How Pain Has Interfered With Your Sleep)
Description: as for outcome 16
Time Frame: Baseline, Weeks 1,2,6,10,14 and Endpoint
Population: ITT population; n = number of participants with data for analysis (n=pregabalin, placebo).
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 148 | 147
score on scale
  Week 1 (n=145,147) | -1.80 (0.18) | -1.12 (0.18)
  Week 2 (n=139,142) | -2.22 (0.22) | -1.86 (0.21)
  Week 6 (n=131,134) | -3.06 (0.21) | -2.68 (0.21)
  Week 10 (n=126,128) | -3.10 (0.22) | -2.71 (0.21)
  Week 14 (n=116,120) | -2.65 (0.23) | -2.90 (0.23)
  Endpoint (n=148,147) | -2.51 (0.22) | -2.74 (0.21)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 1; Test type: Superiority or Other; p = 0.0073, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.68, 95% CI [-1.18 to -0.19], Standard Error of Mean 0.25
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 2; Test type: Superiority or Other; p = 0.2202, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.37, 95% CI [-0.96 to 0.22], Standard Error of Mean 0.30
Statistical Analysis 3: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 6; Test type: Superiority or Other; p = 0.1824, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.39, 95% CI [-0.95 to 0.18], Standard Error of Mean 0.29
Statistical Analysis 4: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 10; Test type: Superiority or Other; p = 0.1872, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.39, 95% CI [-0.98 to 0.19], Standard Error of Mean 0.30
Statistical Analysis 5: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 14; Test type: Superiority or Other; p = 0.4374, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.25, 95% CI [-0.38 to 0.88], Standard Error of Mean 0.32
Statistical Analysis 6: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Endpoint; Test type: Superiority or Other; p = 0.4406, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.23, 95% CI [-0.36 to 0.82], Standard Error of Mean 0.30

26. Secondary Outcome: Change in Brief Pain Inventory-sf Scores (During the Past 24 Hours, How Pain Has Interfered With Your Enjoyment of Life)
Description: as for outcome 16
Time Frame: Baseline, Weeks 1,2,6,10,14 and Endpoint
Population: ITT population; n = number of participants with data for analysis (n=pregabalin, placebo).
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 148 | 146
score on scale
  Week 1 (n=145,146) | -1.52 (0.20) | -1.20 (0.19)
  Week 2 (n=139,141) | -2.20 (0.24) | -2.13 (0.23)
  Week 6 (n=132,131) | -2.69 (0.21) | -2.64 (0.21)
  Week 10 (n=126,127) | -2.59 (0.21) | -2.45 (0.21)
  Week 14 (n=116,119) | -2.78 (0.22) | -2.79 (0.22)
  Endpoint (n=148,146) | -2.64 (0.21) | -2.60 (0.21)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 1; Test type: Superiority or Other; p = 0.2277, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.33, 95% CI [-0.86 to 0.21], Standard Error of Mean 0.27
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 2; Test type: Superiority or Other; p = 0.8407, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.07, 95% CI [-0.71 to 0.58], Standard Error of Mean 0.33
Statistical Analysis 3: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 6; Test type: Superiority or Other; p = 0.8809, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.04, 95% CI [-0.62 to 0.53], Standard Error of Mean 0.29
Statistical Analysis 4: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 10; Test type: Superiority or Other; p = 0.6288, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.14, 95% CI [-0.72 to 0.43], Standard Error of Mean 0.29
Statistical Analysis 5: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Week 14; Test type: Superiority or Other; p = 0.9739, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.01, 95% CI [-0.59 to 0.61], Standard Error of Mean 0.30
Statistical Analysis 6: Comparison: Pregabalin vs Placebo; Table above shows results of statistical analysis for Endpoint; Test type: Superiority or Other; p = 0.8926, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.04, 95% CI [-0.61 to 0.53], Standard Error of Mean 0.29

27. Secondary Outcome: Shift Table NPSI (Neuropathic Pain Symptom Inventory) - Duration of Spontaneous Pain
Description: Number of subjects reporting duration of spontaneous pain. The NPSI includes the temporal item for assessment of duration of spontaneous, ongoing and paroxysmal pain. Assessed using a 5-point specific categorical scale and refers to the past 24 hours at endpoint.
Time Frame: Baseline-Week 14 (Endpoint)
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 128 | 126
participants
  Permanently (baseline&endpoint) | 15 | 21
  Permanently (baseline), 8-12 hours (endpoint) | 11 | 5
  Permanently (baseline), 4-7 hours (endpoint) | 8 | 6
  Permanently (baseline), 1-3 hours (endpoint) | 4 | 5
  Permanently (baseline), < 1 hr (endpoint) | 4 | 5
  8-12 hours (baseline), permanently (endpoint) | 2 | 7
  8-12 hrs (baseline), 8-12 hrs (endpoint) | 10 | 7
  8-12 hrs (baseline), 4-7 hrs (endpoint) | 5 | 9
  8-12 hrs (baseline), 1-3 hours (endpoint) | 4 | 4
  8-12 hrs (baseline), <1 hr (endpoint) | 8 | 5
  4-7 hrs (baseline), permanently (endpoint) | 3 | 3
  4-7 hrs (baseline), 8-12 hrs (endpoint) | 7 | 6
  4-7 hrs (baseline), 4-7 hrs (endpoint) | 9 | 9
  4-7 hrs (baseline), 1-3 hrs (endpoint) | 3 | 8
  4-7 hrs (baseline), < 1 hr (endpoint) | 7 | 8
  1-3 hrs (baseline), permanently (endpoint) | 1 | 0
  1-3 hrs (baseline), 8-12 hrs (endpoint) | 2 | 2
  1-3 hrs (baseline), 4-7 hrs (endpoint) | 1 | 5
  1-3 hrs (baseline), 1-3 hrs (endpoint) | 6 | 3
  1-3 hrs (baseline), <1 hr (endpoint) | 9 | 5
  Less than 1 hr (baseline), permanently (endpoint) | 0 | 1
  Less than 1 hr (baseline), 8-12 hrs (endpoint) | 2 | 0
  Less than 1 hr (baseline), 4-7 hrs (endpoint) | 0 | 0
  Less than 1 hr (baseline), 1-3 hrs (endpoint) | 1 | 2
  <1 hr (baseline), <1 hr (endpoint) | 6 | 0

28. Secondary Outcome: Shift Table in NPSI (Neuropathic Pain Symptom Inventory)- Number of Pain Attacks
Description: Number of subjects reporting pain attacks. The NPSI includes the temporal item for assessing the numbers of pain attacks. Assessed using a 5-point specific categorical scale and refers to the past 24 hours at endpoint.
Time Frame: Baseline-Week 14 (Endpoint)
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 119 | 119
participants
  >20 attacks (baseline & endpoint) | 4 | 6
  >20 attacks (baseline), 11-20 attacks (endpoint) | 2 | 4
  >20 attacks (baseline), 6-10 attacks (endpoint) | 1 | 4
  >20 attacks (baseline), 1-5 attacks (endpoint) | 3 | 3
  >20 attacks (baseline), no pain attacks (endpoint) | 3 | 2
  11-20 attacks (baseline), >20 attacks (endpoint) | 2 | 0
  11-20 attacks (baseline), 11-20 attacks (endpoint) | 2 | 2
  11-20 attacks (baseline), 6-10 attacks (endpoint) | 7 | 8
  11-20 attacks (baseline), 1-5 attacks (endpoint) | 10 | 8
  11-20 attacks (baseline), no attacks (endpoint) | 9 | 5
  6-10 attacks (baseline), >20 attacks (endpoint) | 1 | 7
  6-10 attacks (baseline), 11-20 attacks (endpoint) | 2 | 2
  6-10 attacks (baseline), 6-10 attacks (endpoint) | 5 | 8
  6-10 attacks (baseline), 1-5 attacks (endpoint) | 14 | 17
  6-10 attacks (baseline), no attacks (endpoint) | 6 | 4
  1-5 attacks (baseline), >20 attacks (endpoint) | 3 | 1
  1-5 attacks (baseline), 11-20 attacks (endpoint) | 3 | 2
  1-5 attacks (baseline), 6-10 attacks (endpoint) | 7 | 3
  1-5 attacks (baseline), 1-5 attacks (endpoint) | 21 | 15
  1-5 attacks (baseline), no attacks (endpoint) | 10 | 11
  no attacks (baseline), >20 attacks (endpoint) | 0 | 2
  no attacks (baseline), 11-20 attacks (endpoint) | 0 | 0
  no attacks (baseline), 6-10 attacks (endpoint) | 0 | 1
  no attacks (baseline), 1-5 attacks (endpoint) | 1 | 3
  no attacks (baseline), no attacks (endpoint) | 3 | 1

29. Secondary Outcome: Change in Number of Pain Attacks Compared to Baseline - NPSI (Neuropathic Pain Symptom Inventory)
Description: Change from baseline in the number of pain attacks at endpoint. The NPSI includes the temporal item for assessing the numbers of pain attacks. Assessed using a 5-point specific categorical scale and refers to the past 24 hours at endpoint.
Time Frame: Baseline, Week 14
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 119 | 119
participants
  Improved from baseline to endpoint | 65 | 66
  No change from baseline to endpoint | 35 | 32
  Worsened from baseline to endpoint | 19 | 21
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.7136, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]

30. Secondary Outcome: Duration of Spontaneous Pain-NPSI (Neuropathic Pain Symptom Inventory)
Description: Change from baseline to endpoint in the duration of spontaneous pain. The NPSI includes the temporal item for assessment of duration of spontaneous, ongoing and paroxysmal pain. Assessed using a 5-point specific categorical scale and refers to the past 24 hours at endpoint.
Time Frame: Baseline, Week 14
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 128 | 126
participants
  Improved from baseline to endpoint | 63 | 60
  No change from baseline to endpoint | 46 | 40
  Worsened from baseline to endpoint | 19 | 26
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.6729, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]

31. Secondary Outcome: Gracely Pain Scale Score
Description: The modified Gracely Pain Scale is a 13-point verbal rating scale based on sensory pain descriptors ranked by severity from nothing (rank = 0) to extremely intense (rank = 15). Subjects selected the verbal descriptors that best matched their average neuropathic pain during the last 24 hours prior to assessment.
Time Frame: Week 14
Population: ITT Population
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 128 | 127
score on scale | -2.70 (3.36) | -2.76 (3.19)

32. Secondary Outcome: Quantitative Assessments of Neuropathic Pain (QANeP) Maximum Sensory Thresholds : Shift Table
Description: Shift from baseline in maximum sensory thresholds (in grams representing the force equivalent of various sizes of von Frey filaments) as measured on QANeP. Improved - decrease in the maximum of the 3 trials at endpoint. Worsened - an increase. Note:Sensory Thresholds are the highest values of the 3 trials at baseline (Week=0) and endpoint (Week 14)
Time Frame: Baseline-Week 14 (Endpoint)
Population: ITT Population; Pregabalin weight range- 3.61, 4.31, 4.56, 5.07, 6.65 and not perceived. Placebo weight range- 2.83, 3.61, 4.31, 4.56, 5.07, 6.65 and not perceived
Measure: Number; unit: participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 149 | 150
participants
  Weight 2.83 Improved | 0 | 0
  Weight 2.83 No Change | 0 | 1
  Weight 2.83 Worsened | 0 | 3
  Weight 3.61 Improved | 1 | 2
  Weight 3.61 No Change | 3 | 2
  Weight 3.61 Worsened | 9 | 4
  Weight 4.31 Improved | 4 | 12
  Weight 4.31 No Change | 17 | 13
  Weight 4.31 Worsened | 8 | 18
  Weight 4.56 Improved | 5 | 6
  Weight 4.56 No Change | 4 | 7
  Weight 4.56 Worsened | 9 | 8
  Weight 5.07 Improved | 10 | 15
  Weight 5.07 No Change | 8 | 3
  Weight 5.07 Worsened | 10 | 5
  Weight 6.65 Improved | 12 | 5
  Weight 6.65 No Change | 7 | 6
  Weight 6.65 Worsened | 2 | 0
  Not Perceived Improved | 3 | 4
  Not Perceived No Change | 8 | 5
  Not Perceived Worsened | 0 | 0

33. Secondary Outcome: Quantitative Assessments of Neuropathic Pain (QANeP) Median Sensory Thresholds : Shift Table
Description: Shift from baseline in median sensory thresholds (designated as Weight) from 3 trials as measured on the QANeP. Improved - a decrease in the median of the three trials at endpoint. Worsened - an increase. Note: Sensory Thresholds are the highest values of the three Trials at both baseline (Week=0) and endpoint (Week 14).
Time Frame: Baseline-Week 14 (Endpoint)
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 149 | 150
participants
  Weight 2.83 Improved | 0 | 0
  Weight 2.83 No Change | 1 | 3
  Weight 2.83 Worsened | 5 | 3
  Weight 3.61 Improved | 0 | 2
  Weight 3.61 No Change | 10 | 9
  Weight 3.61 Worsened | 10 | 13
  Weight 4.31 Improved | 12 | 11
  Weight 4.31 No Change | 7 | 11
  Weight 4.31 Worsened | 9 | 12
  Weight 4.56 Improved | 8 | 7
  Weight 4.56 No Change | 6 | 8
  Weight 4.56 Worsened | 5 | 7
  Weight 5.07 Improved | 16 | 11
  Weight 5.07 No Change | 5 | 3
  Weight 5.07 Worsened | 6 | 1
  Weight 6.65 Improved | 10 | 8
  Weight 6.65 No Change | 2 | 3
  Weight 6.65 Worsened | 0 | 0
  Not Perceived Improved | 2 | 3
  Not Perceived No Change | 6 | 4
  Not Perceived Worsened | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential info other than study results.